CLINICAL TRIAL: NCT05978323
Title: The Effect of Brief Interventıon on Behavıoral Change, Anthropometrıc and Metabolıc Varıables In Overweıght Women wıth Low Health Lıteracy
Brief Title: The Effect of a Brief Intervention on Behavıoral Change, Anthropometric and Metabolic Variables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Yasemin Guven, Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MeU-YGUVEN-001
Record Dates: First submitted 2023-07-02; First posted 2023-08-07 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Brief Intervention
Keywords: Brief intervention; Overweight; Health literacy; Weight change; Metabolic variables
MeSH Terms: conditions — Overweight; Body Weight Changes | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Prospective, parallel randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: For each group, 21 blocks were created by generating random numbers in Excel by a person other than the researcher and assigned to groups A and B. The assignment of the intervention and control groups was made by drawing lots. Index cards prepared for two primary healthcare organizations by block randomization by the researcher who did not participate in the clinical part of the study will be placed in closed opaque envelopes and their sequence numbers will be written on the envelopes. The research data will be entered into the computer database by the researcher as coded as A and B. Statistical analyses will be performed by the researcher who did not participate in the data collection phase according to this code. The research report will also be written in coded form. Research participants and statistical evaluators were planned to be blind to group assignment, single-blind, and statistician blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief intervention (Experimental): Intervention Group: Short face-to-face intervention interviews will be conducted with individuals in the intervention group. Interviews will be held in primary healthcare organizations' meeting rooms. Brief intervention interviews will be conducted with the intervention group. It was determined as the first evaluation and the follow-ups on the 1st day, 15th day, 1st month, 3rd month, and the last evaluation (6th month). Brief interventions, 5A for those who are ready to change their behavior (Ask, Advise, Assess, Assist, Arrange); Those who are not ready to change their behavior 5R (Relevance, Risks, Rewards, Roadblocks, Repetition) model will be used. Brief intervention interviews will take an average of 20-30 minutes. The talks will include awareness of overweight and obesity, a healthy diet, and exercise. By the researcher's prepared will be used for individuals with low health literacy educational materials.
  Interventions: Behavioral: Brief intervention
- Control (No Intervention): The control group will not be intervened except for the first and last face-to-face evaluation. At the end of the research, training materials for weight loss will be given.

INTERVENTIONS:
Behavioral: Brief intervention — Short face-to-face intervention interviews will be conducted with individuals in the intervention group. Interviews will be held in primary healthcare organizations' meeting rooms. Brief intervention interviews will be conducted with the intervention group. It was determined as the first evaluation and the follow-ups on the 1st day, 15th day, 1st month, 3rd month, and the last evaluation (6th month). Brief interventions, 5A for those who are ready to change their behavior (Ask, Advise, Assess, Assist, Arrange); Those who are not ready to change their behavior 5R (Relevance, Risks, Rewards, Roadblocks, Repetition) model will be used. Brief intervention interviews will take an average of 20-30 minutes. The talks will include awareness of overweight and obesity, a healthy diet, and exercise. By the researcher's prepared will be used for individuals with low health literacy educational materials.
  Arms: Brief intervention

SUMMARY:
This study will evaluate the effect of a brief intervention on anthropometric and metabolic changes in overweight women with low health literacy. The total number of samples was determined as 88. It was decided to recruit a total of 124 people, 62 people in each group, with a 40% loss in the groups. Brief intervention interviews will be conducted with the intervention group. Brief intervention interviews will take an average of 20-30 minutes and four times. The control group will not be intervened except for the first and last evaluations.

DETAILED DESCRIPTION:
This study will evaluate the effect of a brief intervention on anthropometric and metabolic changes in overweight women with low health literacy. The total number of samples was determined as 88, 44 in each of the intervention and control groups. It was decided to recruit a total of 124 people, 62 people in each group, with a 40% loss in the groups. Randomization will be performed after obtaining consent from the participants who meet the eligibility and exclusion criteria. The sampled individuals will be assigned to the Intervention and Control groups according to the block randomization method. Brief intervention interviews will be conducted with the intervention group. It was determined as the first evaluation and the follow-ups on the 1st day, 15th day, 1st month, 3rd month, and the last evaluation (6th month). Brief interventions, 5A for those who are ready to change their behavior (Ask, Advise, Assess, Assist, Arrange); those who are not ready to change their behavior 5R (Relevance, Risks, Rewards, Roadblocks, Repetition) model will be used. At the end of brief interventions applied to overweight women with low health literacy for 20-30 minutes, a total of four times; weight change, waist circumference change, blood pressure change, blood glucose change, blood lipid change, diet, and exercise behaviors will be evaluated. The control group will not be intervened except for the first and last evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Having heart disease, stroke, and chronic kidney failure diagnosed by a physician,
* Having diabetes that requires the use of insulin,
* Having hypothyroidism that prevents weight loss,
* Participating in a weight management program in the last 3 months,
* Being diagnosed with a disease that causes deterioration in cognitive processes such as Alzheimer's and dementia,
* Having a diagnosed physical or neurological problem that prevents him from doing physical activity,
* People who plan to become pregnant or become pregnant during the trial period (8 months after enrollment in the trial)

Exclusion Criteria:

* Between 12.09.2023 and 24.06.2024 two Primary healthcare organization applied,
* Volunteered to participate in the research,
* Women between the ages of 30-65,
* The level of health literacy is limited-restricted,
* 25≥ BMI < 30,
* Those who can read and understand Turkish will be included in the study.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of weight change | Change from before implementation three and six months of practice.
  The weight will be evaluated by measuring the weight.

SECONDARY OUTCOMES:
The exercise habits will be evaluated using the Exercise Behavior Change Model Scales. | Change from before implementation and six months of practice.
  The highest score that can be obtained from the scale is 140, and the lowest score is 28. The higher the scale score indicates that the individual's chance of being successful in change increases.
The eating habits will be evaluated using the Nutrition Processes of Change Scale. | Change from before implementation and six months of practice.
  The highest score that can be obtained from the scale is 240, and the lowest score is 48. Higher scores from the scale indicate more positive values for change.
The Mediterranean diet will be evaluated using the Mediterranean Diet Adherence Screener (MEDAS). | Change from before implementation and six months of practice.
  A total score of 7 and 8 on the scale indicates an acceptable degree of adherence to the Mediterranean diet, and a score of 9 and above indicates strict adherence to the Mediterranean diet.
Waist circumference measurement and evaluation | Change from before implementation, three and six months of practice.
  Waist circumference will be measured by the researcher with a tape measure from the thinnest part of the waist at the level of the navel, passing through the anterior superior of the spina iliaca. Waist circumference <80 will be considered "low risk", >80-88 will be considered "high risk" and >88 will be considered "very high risk."
Measurement and evaluation of blood pressure (BP) | Change from before implementation, three and six months of practice.
  By the Hypertension Diagnosis and Treatment Guidelines, measures will be made on both arms, and the average will be recorded. BP below 120/80 mmHg is normal, mean systolic BP of 120-139 mmHg and/or mean diastolic BP of 80-89 mmHg increased, and mean systolic BP ≥140 mmHg and/or mean diastolic BP ≥90 mmHg will be considered hypertension.
Evaluation of fasting plasma glucose level | Change from before implementation and six months of practice.
  "Fasting plasma glucose" ≥ 126 mg/dl or "suspected diabetes mellitus" if values of "200 mg/dl" and above in a random measurement area will be evaluated as.
Evaluation of glycosylated hemoglobin A1c (HbA1c) level | Change from before implementation and six months of practice.
  A1c 5.7-6.4% (39-47 mmol/mol) will be considered a "high-risk group." A1c ≥6.5% (≥48 mmol/mol) will be considered as "diabetes mellitus."
Evaluation of blood lipid changes (Total cholesterol, HDL, LDL cholesterol, and triglyceride level) | Change from before implementation and six months of practice.
  Total cholesterol <200 mg/dL is considered "optimal," 200-239 mg/dL is "borderline high" and >240 mg/dL is "high". will be evaluated.
  HDL cholesterol ≥60 mg/dL will be considered "optimal", 50-59 mg/dL will be considered "borderline high" and <50 mg/dL will be considered "high."
  LDL cholesterol <100 mg/dL will be considered "optimal", 100-129 mg/dL will be considered "normal," 130-159 mg/dL will be considered "borderline high" and ≥160-189 mg/dL will be considered ''high,'' ≥190 mg/dL will be considered "very high."
  A triglyceride of <150 mg/dL will be considered "normal,"150-199 mg/dL will be considered "borderline high," 200-500 mg/dL will be considered "high" and ≥500 mg/dL will be considered "very high."
Body mass index (BMI) evaluation | Change from before implementation, three and six months of practice.
  BMI <18.5-24.9 kg/m2 will be defined as "normal", BMI between 25-29.9 kg/m2 will be defined as "overweight", and BMI≥ 30 kg/m2 will be defined as "obese".

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Güven, Master, Principal Investigator — Mersin University
Locations (1):
- Turkey, Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR